CLINICAL TRIAL: NCT01551836
Title: A Randomised, Two Way Crossover Study to Determine the Time at Which Therapeutic Plasma Concentrations of Paracetamol Are Achieved in Two Marketed Formulations
Brief Title: At What Time Therapeutic Plasma Concentrations of Paracetamol Are Achieved in Two Marketed Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: E3870651
Record Dates: First submitted 2011-06-23; First posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Healthy Volunteer
Keywords: pharmacokinetics; paracetamol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol formulation 1 (Other): Higher dose level of marketed paracetamol (compared to the other dosage arm)
  Interventions: Drug: Paracetamol formulation 1
- Paracetamol formulation 2 (Other): Lower paracetamol concentrations
  Interventions: Drug: Paracetamol formulation 2

INTERVENTIONS:
Drug: Paracetamol formulation 1 — formulation 1
  Arms: Paracetamol formulation 1
Drug: Paracetamol formulation 2 — Formulation 2
  Arms: Paracetamol formulation 2

SUMMARY:
This will be a single centre, open label, randomised, two-way crossover study in healthy volunteers under semi-fed conditions. Two formulations of paracetamol, are being tested in this study to establish at what time point a therapeutic concentration of paracetamol in the blood is reached. Subjects will attend a screening visit to check if they are eligible for study participation then within 15 days they will check-in to the unit for a stay of approximately 48 hours (hrs). They will be given a single dose of one of the preparations on the first day and then the other preparation on the next day. Regular blood samples will be taken along with other assessments for safety.

ELIGIBILITY:
Inclusion Criteria:

* Males in good general heatlh and Body Mass Index between 19-28 kg/m2

Exclusion Criteria:

* Disease

  1. Current liver impairment, renal impairment, history of or active gastrointestinal ulcers, uncontrolled hypertension, haemophilia or other bleeding disorders.
  2. Current or recurrent disease, within 12 months of the screening, that could affect the action, absorption or disposition of the study formulations or clinical or laboratory assessments (e.g. hepatic disorders, renal insufficiency, congestive heart failure).
  3. Current or relevant previous history, within 12 months of the screening visit, of serious, severe or unstable physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study treatments or procedures.
* Medications

  1. Current or regular use at screening of any prescription, herbal or Over the Counter (OTC) medication including paracetamol, aspirin, metaclopramide, domperidone, cholestyramine, angiotensin -converting enzyme (ACE) inhibitors, acetazolamide, anticonvulsants, diuretics, methotrexate, non-steroidal anti-inflammatory drugs (NSAIDs) and oral hypoglycemics within the past 48 hrs and monoamine oxidase inhibitors, tricyclic antidepressants, beta blockers and anticoagulants such as warfarin and heparin within the past 2 weeks.
  2. Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to the screening visit (some examples of inducers: barbiturates, theophylline; inhibitors: cimetidine, erythromycin).
  3. Subjects for whom the use of any of the study drugs is contraindicated.
* Virology Screening Positive screening for serum Hepatitis B surface antigen, Hepatitis C antibodies or human immunodeficiency virus (HIV).
* Drug Screen

  1. Positive urine screen for drugs of abuse at screening and/or Day-1.
  2. Positive alcohol breath test on Day-1.
* Smoking

  1. Smoking more than five cigarettes a day.
  2. Prior (within 7 days of dosing on Day 1) or current use of any other nicotine containing products, other than cigarettes/pipes/cigars.
* Blood donation Has donated blood or plasma or any other blood product within 3 months of the screening visit. Subjects for whom participation in this study would result in having donated more than 1500 ml of blood within the previous 12 months.
* Nutrition

  1. Is a vegetarian or is under a sodium restricted diet.
  2. Has consumed poppy seed containing foods within 3 days prior to the screening visit and admission on Day -1.
  3. Has consumed food and beverages containing grapefruit, Seville oranges or marmalade within 24 hrs prior to admission on Day -1.
  4. Has consumed caffeine containing drinks or food (e.g. tea, coffee, chocolate and cola) 24 hrs prior to admission on Day -1.
  5. Has consumed alcohol 36 hrs prior to admission on Day -1.
* Has undertaken any unusually strenuous physical activity 24 hrs prior to the screening visit or check-in on Day 1.
* Weight Weight below 50 kg.
* Haemoglobin Subjects with haemoglobin level below 12.0 gram /decilitre (dl).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Mean time to therapeutic levels of plasma concentration | within a single day

SECONDARY OUTCOMES:
Mean plasma concentrations | within a single day

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Belfast, Northern Ireland, United Kingdom